CLINICAL TRIAL: NCT00792285
Title: Automated Telephone Outreach With Speech Recognition to Improve Colorectal Cancer Screening: A Randomized Controlled Trial
Brief Title: RCT of Automated Telephone Outreach to Improve Colorectal Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Pilgrim Health Care (Other)
Responsible Party: Steven R. Simon, MD / Principal Investigator, Harvard Pilgrim Health Care
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ATO-SR CRC
Record Dates: First submitted 2008-11-13; First posted 2008-11-17 (Estimated); Last update posted 2008-11-17 (Estimated); Status verified 2008-11

CONDITIONS: Colorectal Cancer
Keywords: Colon cancer; Prevention; Screening; Telephone
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Automated Telephone Outreach (Experimental): Automated Telephone Outreach with Speech Recognition
  Interventions: Behavioral: Automated Telephone Outreach with Speech Recognition
- Usual Care (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: Automated Telephone Outreach with Speech Recognition — Automated Telephone Outreach with Speech Recognition calls to health plan members to promote screening
  Arms: Automated Telephone Outreach

SUMMARY:
This large randomized controlled trial is testing the effectiveness of automated telephone outreach with speech recognition to improve rates of screening for colorectal cancer. The hypothesis is that the intervention improves rates of screening overall and specifically rates of colonoscopy.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the second leading cause of cancer-related mortality in the United States. Despite widespread dissemination of evidence-based guidelines recommending CRC screening, a large proportion of eligible individuals do not undergo screening. A variety of interventions have been tested to increase screening in primary care, but there remains an urgent imperative to develop and evaluate cost-effective and widely applicable approaches to promoting screening. In March 2005, Harvard Pilgrim Health Care, a large non-profit HMO in New England, carried out an internally funded program to increase CRC screening. The HMO randomized 80,000 members aged 50 to 64 years to receive automated telephone outreach with speech recognition or usual care. The intervention entailed the telephone engagement of members in a dialogue with a computer-programmed, responsive human voice about the importance of CRC screening, the options for undergoing screening, and encouragement to follow-up with their primary care physicians. The present study involves a 12-month follow-up of all eligible members randomized to intervention or usual care in March 2005, with assessment of the effect of the intervention on rates of CRC screening. This study has important implications for increasing CRC screening. With health plans expanding efforts to screen large populations for CRC and other malignancies, automated telephone outreach with speech recognition can reach large numbers of individuals with educational and reminder messages. It is important to know whether these efforts to promote screening are effective in overcoming known disparities in screening for CRC. If proven effective and cost-effective, this technology has the potential for widespread adoption and population-wide improvements in CRC screening and other prevention-related behaviors, with the ultimate public health goal of reducing the burden of suffering attributable to cancer and its complications.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-64 at baseline
* Continuous enrollment in health plan

Exclusion Criteria:

* Prior request for exclusion from research or quality improvement
* No telephone number on file
* Enrolled in other telephone-based outreach program of the health plan
* Share household with another eligible member
* Evidence of colorectal cancer or polyps at baseline
* Evidence of prior screening at baseline such that screening is not due at time of intervention

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80000 (Actual)
Dates: Start 2005-03; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
colorectal cancer screening | one year

SECONDARY OUTCOMES:
colonoscopy screening | one year

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Simon, MD, Principal Investigator — Harvard Pilgrim Health Care
Locations (1):
- Harvard Pilgrim Health Care, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Simon SR, Zhang F, Soumerai SB, Ensroth A, Bernstein L, Fletcher RH, Ross-Degnan D. Failure of automated telephone outreach with speech recognition to improve colorectal cancer screening: a randomized controlled trial. Arch Intern Med. 2010 Feb 8;170(3):264-70. doi: 10.1001/archinternmed.2009.522. PMID 20142572